CLINICAL TRIAL: NCT00221923
Title: African Descent and Glaucoma Evaluation Study (Formerly African Americans With Glaucoma Study)
Brief Title: African Descent and Glaucoma Evaluation Study
Acronym: ADAGES
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of California, San Diego (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Linda Zangwill, Principal Investigator, University of California, San Diego
Other Study IDs: NEI U10 EY 14267; R01EY023704 (NIH); R01EY026574 (NIH)
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Primary Open Angle Glaucoma
Keywords: Primary open angle glaucoma; African American; Glaucoma/pathology; Glaucoma/ physiopathology; Nerve Fibers/pathology; Risk factor glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy individuals: They will be considered if they are above 30 years old. There is no upper age limit. Subject can be either male or female, and from African or European Descent. They must speak, read, and understand English. They can be diagnosed with other health disorders.
- Persons at risk for or with primary open angle glaucoma: They will be considered if they are above 30 years old. There is no upper age limit. Subject can be either male or female, and from African or European Descent. They must speak, read, and understand English. They can be diagnosed with other health disorders.

SUMMARY:
According to the National Eye Institute, Glaucoma affects about three million Americans. Among Blacks in the United States, open- angle glaucoma is the leading cause of irreversible visual loss. Glaucoma is four times more likely to develop in Blacks than in Whites.

This is a prospective longitudinal, multi- site observational cohort study designed to obtain visual function and optic nerve structure data on eyes of Black and White Americans. The investigators will evaluate the relationship between changes in the structure of the eye and the vision loss caused by glaucoma.This is the first study where both populations are matched for quality of care and equal access to care.

DETAILED DESCRIPTION:
The purpose of the study is:

1. To further determine the nature of vision loss and optic nerve structural change associated with glaucoma. Using recently developed measures of visual function and techniques for imaging the eye, we will use a multivariate approach for analysis of the functional and structural changes associated with glaucoma to delineate further the relationship of these changes to the underlying physiological mechanisms..
2. To evaluate and improve new diagnostic and monitoring techniques encompassing measures of visual function and optic nerve and retina nerve fiber layer structure and to compare the rate and patterns of progression of glaucomatous damage in Black and White eyes.
3. To improve techniques for evaluation of current management and new therapies for glaucoma as they become available. We will expand our analysis using multivariate techniques incorporating visual function, optic nerve structure, and various risk factors to improve detection of true change. We will determine whether the benefits found in Whites using visual function specific perimetry and optic disc imaging for earlier detection and for monitoring progression are also found for Blacks.
4. To determine the quantitative temporal relationships between recognizable optic nerve damage and measurable visual field loss and how these relationships differ among Black and White patients. Using new techniques with improved sensitivity, the detection and monitoring of early optic disc defects may provide profiles of people at risk for developing glaucomatous visual function loss thus better defining target populations for treatment.

ELIGIBILITY:
Inclusion Criteria:

* Open angles
* Best-corrected acuity of 20/40 or better
* Spherical refraction within + 5.0 D, and cylinder within + 3.0 D with plus OR minus cylinders
* ≥ 18 years old
* A family history of glaucoma is allowed
* Ability to obtain adequate or better quality stereophotographs
* Ability to do reliable standard Humphrey 30-2 or 24-2 visual fields
* Participants with glaucoma or at risk for glaucoma or healthy controls

Exclusion Criteria:

* History of intraocular surgery (except uncomplicated cataract or glaucoma surgery)
* Problems other than Glaucoma affecting color vision
* Non glaucomatous secondary causes of elevated IOP ( e.g. iridocyclitis, trauma)
* Other intraocular eye disease
* Other diseases affecting visual field (e:g pituitary lesions, demyelinating diseases, HIV+ or AIDS, or diabetic retinopathy) with medications known to affect visual field sensitivity
* Problems other than Glaucoma affecting color vision

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults of African or European descent based on self-report.
Sampling Method: Non-Probability Sample
Enrollment: 1540 (Estimated)
Dates: Start 2002-09 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Linda M Zangwill, Ph.D., Principal Investigator — University of California, San Diego
Locations (3):
- United States (3):
  - University of Alabama-Callahan Eye Foundation, Prof. Bldg., Birmingham, Alabama
  - UCSD Hamilton Glaucoma Center, La Jolla, California
  - New York Eye & Ear Infirmary, New York, New York

REFERENCES:
- [Background] Sample PA, Bosworth CF, Blumenthal EZ, Girkin C, Weinreb RN. Visual function-specific perimetry for indirect comparison of different ganglion cell populations in glaucoma. Invest Ophthalmol Vis Sci. 2000 Jun;41(7):1783-90. PMID 10845599
- [Background] Racette L, Boden C, Kleinhandler SL, Girkin CA, Liebmann JM, Zangwill LM, Medeiros FA, Bowd C, Weinreb RN, Wilson MR, Sample PA. Differences in visual function and optic nerve structure between healthy eyes of blacks and whites. Arch Ophthalmol. 2005 Nov;123(11):1547-53. doi: 10.1001/archopht.123.11.1547. PMID 16286617
- [Background] Bathija R, Zangwill L, Berry CC, Sample PA, Weinreb RN. Detection of early glaucomatous structural damage with confocal scanning laser tomography. J Glaucoma. 1998 Apr;7(2):121-7. PMID 9559499
- [Background] Zangwill L, Knauer S, Williams JM, Weinreb RN, Retinal fiber layer assessment by scanning laser polarimetery, optical coherence tomography and retinal nerve fiber layer photography. In: Lemij HG, Schuman JS, eds. The Shape of Glaucoma, Quantitative Neural Imaging Techniques. The Hague Kugler Publications, 2000:239-252
- [Background] Wilson MR. Glaucoma in blacks: where do we go from here? JAMA. 1989 Jan 13;261(2):281-2. No abstract available. PMID 2909027
- [Background] Munoz B, West SK, Rubin GS, Schein OD, Quigley HA, Bressler SB, Bandeen-Roche K. Causes of blindness and visual impairment in a population of older Americans: The Salisbury Eye Evaluation Study. Arch Ophthalmol. 2000 Jun;118(6):819-25. doi: 10.1001/archopht.118.6.819. PMID 10865321
- [Background] Tielsch JM, Sommer A, Katz J, Royall RM, Quigley HA, Javitt J. Racial variations in the prevalence of primary open-angle glaucoma. The Baltimore Eye Survey. JAMA. 1991 Jul 17;266(3):369-74. PMID 2056646
- [Background] Javitt JC, McBean AM, Nicholson GA, Babish JD, Warren JL, Krakauer H. Undertreatment of glaucoma among black Americans. N Engl J Med. 1991 Nov 14;325(20):1418-22. doi: 10.1056/NEJM199111143252005. PMID 1922253
- [Background] Sample PA, Weinreb RN, Boynton RM. Acquired dyschromatopsia in glaucoma. Surv Ophthalmol. 1986 Jul-Aug;31(1):54-64. doi: 10.1016/0039-6257(86)90051-2. PMID 3529468
- [Background] Sample PA, Weinreb RN. Color perimetry for assessment of primary open-angle glaucoma. Invest Ophthalmol Vis Sci. 1990 Sep;31(9):1869-75. PMID 2211033
- [Background] Sample PA, Madrid ME, Weinreb RN. Evidence for a variety of functional defects in glaucoma-suspect eyes. J Glaucoma. 1994 Summer;3 Suppl 1:S5-18. PMID 19920588
- [Background] Sample PA, Johnson CA, Haegerstrom-Portnoy G, Adams AJ. Optimum parameters for short-wavelength automated perimetry. J Glaucoma. 1996 Dec;5(6):375-83. PMID 8946293
- [Background] Yamagishi N, Anton A, Sample PA, Zangwill L, Lopez A, Weinreb RN. Mapping structural damage of the optic disk to visual field defect in glaucoma. Am J Ophthalmol. 1997 May;123(5):667-76. doi: 10.1016/s0002-9394(14)71079-7. PMID 9152072
- [Background] Anton A, Yamagishi N, Zangwill L, Sample PA, Weinreb RN. Mapping structural to functional damage in glaucoma with standard automated perimetry and confocal scanning laser ophthalmoscopy. Am J Ophthalmol. 1998 Apr;125(4):436-46. doi: 10.1016/s0002-9394(99)80183-4. PMID 9559728
- [Background] Girkin CA, Emdadi A, Sample PA, Blumenthal EZ, Lee AC, Zangwill LM, Weinreb RN. Short-wavelength automated perimetry and standard perimetry in the detection of progressive optic disc cupping. Arch Ophthalmol. 2000 Sep;118(9):1231-6. doi: 10.1001/archopht.118.9.1231. PMID 10980768
- [Background] Sample PA. What does functional testing tell us about optic nerve damage? Surv Ophthalmol. 2001 May;45 Suppl 3:S319-24; discussion S332-4. doi: 10.1016/s0039-6257(01)00196-5. PMID 11377456
- [Background] Bowd C, Zangwill LM, Berry CC, Blumenthal EZ, Vasile C, Sanchez-Galeana C, Bosworth CF, Sample PA, Weinreb RN. Detecting early glaucoma by assessment of retinal nerve fiber layer thickness and visual function. Invest Ophthalmol Vis Sci. 2001 Aug;42(9):1993-2003. PMID 11481263
- [Background] Goldbaum MH, Sample PA, Chan K, Williams J, Lee TW, Blumenthal E, Girkin CA, Zangwill LM, Bowd C, Sejnowski T, Weinreb RN. Comparing machine learning classifiers for diagnosing glaucoma from standard automated perimetry. Invest Ophthalmol Vis Sci. 2002 Jan;43(1):162-9. PMID 11773027
- [Background] Johnson CA, Sample PA, Cioffi GA, Liebmann JR, Weinreb RN. Structure and function evaluation (SAFE): I. criteria for glaucomatous visual field loss using standard automated perimetry (SAP) and short wavelength automated perimetry (SWAP). Am J Ophthalmol. 2002 Aug;134(2):177-85. doi: 10.1016/s0002-9394(02)01577-5. PMID 12140023
- [Background] Medeiros FA, Sample PA, Weinreb RN. Corneal thickness measurements and visual function abnormalities in ocular hypertensive patients. Am J Ophthalmol. 2003 Feb;135(2):131-7. doi: 10.1016/s0002-9394(02)01886-x. PMID 12566014
- [Background] Racette L, Wilson MR, Zangwill LM, Weinreb RN, Sample PA. Primary open-angle glaucoma in blacks: a review. Surv Ophthalmol. 2003 May-Jun;48(3):295-313. doi: 10.1016/s0039-6257(03)00028-6. PMID 12745004
- [Background] Schiefer U, Flad M, Stumpp F, Malsam A, Paetzold J, Vonthein R, Denk PO, Sample PA. Increased detection rate of glaucomatous visual field damage with locally condensed grids: a comparison between fundus-oriented perimetry and conventional visual field examination. Arch Ophthalmol. 2003 Apr;121(4):458-65. doi: 10.1001/archopht.121.4.458. PMID 12695242
- [Background] Medeiros FA, Sample PA, Weinreb RN. Frequency doubling technology perimetry abnormalities as predictors of glaucomatous visual field loss. Am J Ophthalmol. 2004 May;137(5):863-71. doi: 10.1016/j.ajo.2003.12.009. PMID 15126151
- [Background] Sanchez-Galeana CA, Bowd C, Zangwill LM, Sample PA, Weinreb RN. Short-wavelength automated perimetry results are correlated with optical coherence tomography retinal nerve fiber layer thickness measurements in glaucomatous eyes. Ophthalmology. 2004 Oct;111(10):1866-72. doi: 10.1016/j.ophtha.2004.04.017. PMID 15465548
- [Background] Sample PA, Chan K, Boden C, Lee TW, Blumenthal EZ, Weinreb RN, Bernd A, Pascual J, Hao J, Sejnowski T, Goldbaum MH. Using unsupervised learning with variational bayesian mixture of factor analysis to identify patterns of glaucomatous visual field defects. Invest Ophthalmol Vis Sci. 2004 Aug;45(8):2596-605. doi: 10.1167/iovs.03-0343. PMID 15277482
- [Background] Boden C, Blumenthal EZ, Pascual J, McEwan G, Weinreb RN, Medeiros F, Sample PA. Patterns of glaucomatous visual field progression identified by three progression criteria. Am J Ophthalmol. 2004 Dec;138(6):1029-36. doi: 10.1016/j.ajo.2004.07.003. PMID 15629296
- [Background] Anderson DR. Standard perimetry. Ophthalmol Clin North Am. 2003 Jun;16(2):205-12, vi. doi: 10.1016/s0896-1549(03)00005-1. PMID 12809158
- [Background] Stamper R. L., Sample P. A. and Girkin C. A. (Eds.). (2003). Assessing Visual Function in Clinical Practice. Ophthalmology Clinics of North America, Vol.16, Number . In Anderson J.A and Johnson C.A. (eds.). Frequency-Doubling Technology Perminetry (pp213-226)
- [Background] Stamper R. L., Sample P. A. and Girkin C. A. (Eds.). (2003). Assessing Visual Function in Clinical Practice. Ophthalmology Clinics of North America, Vol.16, Number 2. In Racette L and Sample P.A. (eds.). Short wave automated perimetry. (pp227 -236).
- [Background] Weinreb R.N. and Greve E.L. (Eds.). (2004). Glaucoma diagnosis. Structure and function. The Hague, The Netherlands: Kugler Publications.
- [Derived] Mahmoudinezhad G, Moghimi S, Latif K, Brye N, Walker E, Nishida T, Du KH, Gunasegaran G, Wu JH, Liebmann JM, Fazio MA, Girkin CA, Zangwill LM, Weinreb RN. Number of macula optical coherence tomography scans needed to detect glaucoma progression. Br J Ophthalmol. 2025 May 30;109(6):675-681. doi: 10.1136/bjo-2023-324916. PMID 39663002
- [Derived] Mahmoudinezhad G, Nishida T, Weinreb RN, Baxter SL, Chang AC, Nikkhoy N, Walker E, Liebmann JM, Girkin CA, Moghimi S. Associations of smoking and alcohol consumption with the development of open angle glaucoma: a retrospective cohort study. BMJ Open. 2023 Oct 4;13(10):e072163. doi: 10.1136/bmjopen-2023-072163. PMID 37793935
- [Derived] Bowd C, Belghith A, Rezapour J, Christopher M, Jonas JB, Hyman L, Fazio MA, Weinreb RN, Zangwill LM. Multimodal Deep Learning Classifier for Primary Open Angle Glaucoma Diagnosis Using Wide-Field Optic Nerve Head Cube Scans in Eyes With and Without High Myopia. J Glaucoma. 2023 Oct 1;32(10):841-847. doi: 10.1097/IJG.0000000000002267. Epub 2023 Jul 19. PMID 37523623
- [Derived] Orbach A, Ang GS, Camp AS, Welsbie DS, Medeiros FA, Girkin CA, Fazio MA, Oh WH, Weinreb RN, Zangwill LM, Wu Z. Qualitative Evaluation of the 10-2 and 24-2 Visual Field Tests for Detecting Central Visual Field Abnormalities in Glaucoma. Am J Ophthalmol. 2021 Sep;229:26-33. doi: 10.1016/j.ajo.2021.02.015. Epub 2021 Feb 21. PMID 33626360
- [Derived] Melchior B, De Moraes CG, Paula JS, A Cioffi G, Girkin CA, Fazio MA, N Weinreb R, M Zangwill L, M Liebmann J. Relationship between mean follow-up intraocular pressure, rates of visual field progression and current target intraocular pressure guidelines. Br J Ophthalmol. 2022 Feb;106(2):229-233. doi: 10.1136/bjophthalmol-2020-317406. Epub 2020 Oct 31. PMID 33130556
- [Derived] Wu Z, Medeiros FA, Weinreb RN, Girkin CA, Zangwill LM. Comparing 10-2 and 24-2 Visual Fields for Detecting Progressive Central Visual Loss in Glaucoma Eyes with Early Central Abnormalities. Ophthalmol Glaucoma. 2019 Mar-Apr;2(2):95-102. doi: 10.1016/j.ogla.2019.01.003. Epub 2019 Jan 14. PMID 31742250
- [Derived] Wu Z, Medeiros FA, Weinreb RN, Girkin CA, Zangwill LM. Specificity of various cluster criteria used for the detection of glaucomatous visual field abnormalities. Br J Ophthalmol. 2020 Jun;104(6):822-826. doi: 10.1136/bjophthalmol-2019-314593. Epub 2019 Sep 17. PMID 31530565
- [Derived] De Moraes CG, Hood DC, Thenappan A, Girkin CA, Medeiros FA, Weinreb RN, Zangwill LM, Liebmann JM. 24-2 Visual Fields Miss Central Defects Shown on 10-2 Tests in Glaucoma Suspects, Ocular Hypertensives, and Early Glaucoma. Ophthalmology. 2017 Oct;124(10):1449-1456. doi: 10.1016/j.ophtha.2017.04.021. Epub 2017 May 24. PMID 28551166
- [Derived] Skaat A, De Moraes CG, Bowd C, Sample PA, Girkin CA, Medeiros FA, Ritch R, Weinreb RN, Zangwill LM, Liebmann JM; Diagnostic Innovations in Glaucoma Study and African Descent and Glaucoma Evaluation Study Groups. African Descent and Glaucoma Evaluation Study (ADAGES): Racial Differences in Optic Disc Hemorrhage and Beta-Zone Parapapillary Atrophy. Ophthalmology. 2016 Jul;123(7):1476-83. doi: 10.1016/j.ophtha.2016.03.025. Epub 2016 Apr 23. PMID 27117781
- [Derived] Girkin CA, Nievergelt CM, Kuo JZ, Maihofer AX, Huisingh C, Liebmann JM, Ayyagari R, Weinreb RN, Ritch R, Zangwill LM; ADAGES Study Group. Biogeographic Ancestry in the African Descent and Glaucoma Evaluation Study (ADAGES): Association With Corneal and Optic Nerve Structure. Invest Ophthalmol Vis Sci. 2015 Mar 5;56(3):2043-9. doi: 10.1167/iovs.14-15719. PMID 25744975
- [Derived] Rhodes LA, Huisingh C, Johnstone J, Fazio MA, Smith B, Wang L, Clark M, Downs JC, Owsley C, Girard MJ, Mari JM, Girkin CA. Peripapillary choroidal thickness variation with age and race in normal eyes. Invest Ophthalmol Vis Sci. 2015 Feb 24;56(3):1872-9. doi: 10.1167/iovs.14-16179. PMID 25711640
- [Derived] Hu R, Marin-Franch I, Racette L. Prediction accuracy of a novel dynamic structure-function model for glaucoma progression. Invest Ophthalmol Vis Sci. 2014 Oct 30;55(12):8086-94. doi: 10.1167/iovs.14-14928. PMID 25358735
- [Derived] Tatham AJ, Weinreb RN, Zangwill LM, Liebmann JM, Girkin CA, Medeiros FA. Estimated retinal ganglion cell counts in glaucomatous eyes with localized retinal nerve fiber layer defects. Am J Ophthalmol. 2013 Sep;156(3):578-587.e1. doi: 10.1016/j.ajo.2013.04.015. Epub 2013 Jun 7. PMID 23746612
- [Derived] Tatham AJ, Weinreb RN, Zangwill LM, Liebmann JM, Girkin CA, Medeiros FA. The relationship between cup-to-disc ratio and estimated number of retinal ganglion cells. Invest Ophthalmol Vis Sci. 2013 May 7;54(5):3205-14. doi: 10.1167/iovs.12-11467. PMID 23557744
- [Derived] Bowd C, Lee I, Goldbaum MH, Balasubramanian M, Medeiros FA, Zangwill LM, Girkin CA, Liebmann JM, Weinreb RN. Predicting glaucomatous progression in glaucoma suspect eyes using relevance vector machine classifiers for combined structural and functional measurements. Invest Ophthalmol Vis Sci. 2012 Apr 30;53(4):2382-9. doi: 10.1167/iovs.11-7951. PMID 22427577
- [Derived] Racette L, Liebmann JM, Girkin CA, Zangwill LM, Jain S, Becerra LM, Medeiros FA, Bowd C, Weinreb RN, Boden C, Sample PA; ADAGES Group. African Descent and Glaucoma Evaluation Study (ADAGES): III. Ancestry differences in visual function in healthy eyes. Arch Ophthalmol. 2010 May;128(5):551-9. doi: 10.1001/archophthalmol.2010.58. PMID 20457975
- [Derived] Girkin CA, Sample PA, Liebmann JM, Jain S, Bowd C, Becerra LM, Medeiros FA, Racette L, Dirkes KA, Weinreb RN, Zangwill LM; ADAGES Group. African Descent and Glaucoma Evaluation Study (ADAGES): II. Ancestry differences in optic disc, retinal nerve fiber layer, and macular structure in healthy subjects. Arch Ophthalmol. 2010 May;128(5):541-50. doi: 10.1001/archophthalmol.2010.49. PMID 20457974
- [Derived] Sample PA, Girkin CA, Zangwill LM, Jain S, Racette L, Becerra LM, Weinreb RN, Medeiros FA, Wilson MR, De Leon-Ortega J, Tello C, Bowd C, Liebmann JM; African Descent and Glaucoma Evaluation Study Group. The African Descent and Glaucoma Evaluation Study (ADAGES): design and baseline data. Arch Ophthalmol. 2009 Sep;127(9):1136-45. doi: 10.1001/archophthalmol.2009.187. PMID 19752422
- See also: Website at UCSD — https://shileyeye.ucsd.edu